CLINICAL TRIAL: NCT05969158
Title: An Open, Single-center, Phase II Clinical Study of Hetrombopag in Secondary Prevention of XPO-1 Inhibitor Selinexor Combined With Chemotherapy Induced Thrombocytopenia in Lymphoma
Brief Title: Hetrombopag in Secondary Prevention of XPO-1 Inhibitor-induced Thrombocytopenia in Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-056-01
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Chemotherapy-Induced Thrombocytopenia
MeSH Terms: interventions — hetrombopag

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hetrombopag (Experimental): Hetrombopag 5mg/d
  Interventions: Drug: Hetrombopag

INTERVENTIONS:
Drug: Hetrombopag — After screening, patients who were treated with XPO-1 inhibitor Selinexor combined with chemotherapy and developed chemotherapy-related thrombocytopenia (CIT) after treatment and met the secondary prevention criteria were eligible for inclusion criteria.
  The platelet reduction after the previous chemotherapy was used as the control group:
  The patients did not routinely receive prophylactic platelet elevation therapy after the previous Selinexor combined chemotherapy, and when PLT < 50×109/L.
  Platelet reduction after chemotherapy in secondary prevention unit was used as the experimental group:
  The subjects will initiate treatment with 5 mg hetrombopag once a day, starting orally 5 days before chemotherapy, take it for 5 days (D-5-D-1), and continue taking it orally for 5 days after chemotherapy (D1-D5).
  Other Names: SHR8735

SUMMARY:
To explore the efficacy and safety of hetrombopag for secondary prevention of thrombocytopenia caused by XPO-1 inhibitor Selinexor combined with chemotherapy in patients with lymphoma.

DETAILED DESCRIPTION:
To investigate the efficacy and safety of hetrombopag for secondary prevention of thrombocytopenia in patients with lymphoma treated with XPO-1 inhibitor Selinexor combined with chemotherapy.

ELIGIBILITY:
Inclusion criteria：

1. Age between 18 and 70 years old, gender is not limited;
2. Lymphoma was confirmed by histopathological or cytological examination;
3. The patient needs to receive Selinexor combined chemotherapy containing XPO-1 inhibitor, which may include R-CHOP, R-gemox, DICE, DHAP, SMILE, etc., but is not limited to the above schemes;
4. Patients who do not routinely undergo preventive platelet elevation therapy after the above treatment can receive salvage therapeutic platelet elevation therapy only when the PLT is < 50×109/L;
5. Patients with the lowest platelet value < 50×109/L after the previous course of treatment.
6. The patient's laboratory examination meets the following criteria:

(1) Adequate bone marrow function at Screening: absolute count of blood neutrophils (ANC) ≥1.5×109/L; Platelet (PLT) ≥100×109/L; Hemoglobin (HB) ≥90g/L; (2) Liver function: Without liver metastasis, serum total bilirubin (TBIL) ≤ upper limit of normal (ULN) ×1.5, alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ULN×3; With liver metastasis, TBIL≤ upper limit of normal (ULN) ×3, ALT, AST≤ULN×5; (3) Kidney function: creatinine (Cr) ≤1.5×ULN; (4) Coagulation function: International standardized ratio (INR) of prothrombin time (PT) ≤ULN×1.5;

7. Able to take oral medications;

8. Patients voluntarily sign informed consent;

9. Survival is expected to be ≥12 weeks at the time of screening, and can be treated with the current chemotherapy regimen for at least 2 cycles;

10. Subjects of reproductive age who agree to use reliable contraceptive methods throughout the study period (including male or female condoms, contraceptive foam, contraceptive gel, contraceptive film, contraceptive paste, contraceptive support, abstinence from sex, and insertion of an IUD); Excluding female subjects who have undergone hysterectomy, bilateral salpingectomy, bilateral tubal ligation, or more than 1 year postmenopausal, and male subjects who have undergone bilateral vasectomy or ligation.

Exclusion Criteria:

1. Thrombocytopenia caused by non-tumor chemotherapy drugs, including but not limited to hypersplenism, infection, and bleeding (including severe visceral or intracranial bleeding), occurred within 6 months before screening;
2. A history of blood other than lymphoma and chemotherapy-induced thrombocytopenia (CIT), such as acute lymphoblastic leukemia, acute myeloid leukemia, any myeloid malignancy, myelodysplastic syndrome, myeloproliferative diseases, and multiple myeloma;
3. Any history of arterial or venous thrombosis in the 3 months prior to screening;
4. Patients had clinical manifestations of severe bleeding (such as gastrointestinal bleeding, craniocerebral hemorrhage, etc.) 2 weeks before screening, or previous PLT > 400×109/L;
5. The subject has an allergic reaction to hetrombopag or any of its excipients;
6. Serious cardiovascular disease (such as NYHA heart function) in the 6 months prior to screening Score Ⅲ-Ⅳ), arrhythmias known to increase the risk of thromboembolism, such as atrial fibrillation, after coronary stenting, angioplasty, and coronary artery bypass grafting;
7. The subjects participated in other clinical studies of similar platelet enhancing drugs within 30 days prior to screening;
8. As assessed by the investigator, the subject has any concomitant medical history that could impair the subject's safe completion of the study, such as unstable angina pectoris, renal failure on hemodialysis, or active infection requiring intravenous antibiotics;
9. Subjects who are pregnant or breastfeeding, or who cannot use contraception during the trial;
10. Other circumstances in which the investigator considers the subject unsuitable for participation in the study;
11. HIV infected persons;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-04 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade 3/4 thrombocytopenia during chemotherapy cycles before and after enrollment. | Five days before and five days after chemotherapy
  The incidence of grade 3/4 thrombocytopenia during chemotherapy cycles before and after enrollment.

SECONDARY OUTCOMES:
The minimum and maximum values of median platelets before and after secondary prevention. | 2-3 months
  The minimum and maximum values of median platelets before and after secondary prevention.
The duration of PLT < 75×109 /L, PLT < 50×109 /L and PLT < 25×109 /L before and after chemotherapy; | 2-3 months
  The duration of PLT < 75×109 /L, PLT < 50×109 /L and PLT < 25×109 /L before and after chemotherapy;
The time required for platelet recovery to 100×109/L and 75×109/L; | 2-3 months
  The time required for platelet recovery to 100×109/L and 75×109/L;
The proportion of patients receiving platelet transfusion, the number and amount of transfusion; | 2-3 months
  The proportion of patients receiving platelet transfusion, the number and amount of transfusion;
The proportion of reduced or delayed chemotherapy doses in the next cycle due to thrombocytopenia. | 2-3 months
  The proportion of reduced or delayed chemotherapy doses in the next cycle due to thrombocytopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, MD., Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No